CLINICAL TRIAL: NCT06212466
Title: Magnetocardiography as a Noninvasive Diagnostic Strategy for Suspected Myocardial Ischemia With No Obstructive Coronary Artery Disease
Brief Title: MCG as a Noninvasive Diagnostic Strategy for Suspected INOCA (MICRO2)
Acronym: MICRO2
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MICRO 2.0
Record Dates: First submitted 2023-11-29; First posted 2024-01-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Heart Disease; Coronary Microvascular Disease; Angina; Myocardial Ischemia
Keywords: Magnetocardiography; CardioFlux; Coronary Flow Reserve
MeSH Terms: conditions — Myocardial Ischemia; Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CMD Positive: Patients who have confirmed presence of CMD via invasive angiography/CFR
  Interventions: Device: CardioFlux
- CMD Negative: Patients who have confirmed absence of CMD via invasive angiography/CFR
  Interventions: Device: CardioFlux

INTERVENTIONS:
Device: CardioFlux — The device is a magnetocardiography (MCG) scanner named CardioFlux, which is paired with a cloud processing software for the acquisition, display, and analysis of magnetic fields generated by cardiac electrical activity.

SUMMARY:
A prospective, multicenter, observational, single-arm trial to validate CardioFlux MCG's ability to diagnose myocardial ischemia caused by coronary microvascular dysfunction in patients with suspected ischemia and confirmed no obstructive coronary artery disease (suspected INOCA) by using diagnostic measures of coronary flow reserve (CFR) via invasive angiography as a reference standard for diagnosis.

DETAILED DESCRIPTION:
Magnetocardiography (MCG) is a noninvasive imaging modality that has been extensively studied over the past several decades as a diagnostic imaging solution for various forms of cardiovascular disease. MCG measures the magnetic field that arises from the electrical activity of the heart's pacemaker activity, the very same activity which yields surface electric field potentials as measured by the electrocardiogram. Unlike electrocardiographic signals, however, MCG signals are undistorted by conductive tissue noise, and are highly sensitive to ischemic injury and vortex currents missed by the same electrocardiographic measurements. Accordingly, numerous clinical trials suggest the usefulness of MCG for the evaluation of ischemia in patients with suspected acute coronary syndrome.

There is a growing body of evidence demonstrating the usefulness of MCG in the detection of myocardial ischemia, both in patients with symptoms of ACS, and in patients with stable angina. Since MCG is a functional assessor of depolarization and repolarization heterogeneity, it is hypothesized that MCG may be a useful frontline diagnostic modality to identify CMD in patients who would otherwise have normal coronary CT angiograms and/or stress tests. The proposed study intends to study the diagnostic accuracy of MCG in patients with suspected INOCA.

This demonstrates a significant unmet clinical need in the assessment of patients, and especially women, with INOCA. The current standard of care for these patients is resource/time intensive and associated with a significant rate of non-diagnostic clinical data requiring expensive and invasive evaluation for safe patient management. Magnetocardiography offers the potential for rapid, safe, noninvasive, non-radiologic assessment of the INOCA population, and may lead to earlier treatment strategies for CMD patients.

From the participating clinical sites, patients age ≥18 years who presented with chest pain or exertional dyspnea concerning for myocardial ischemia with no obstructive epicardial CAD on invasive or computed tomographic coronary angiography will be screened and subsequently enrolled when meeting criteria. This is a prospective observational study used for clinical data collection for the clinical validation testing of the CardioFlux MCG system. There will be no intervention introduced by the study device. The interpretation of the CardioFlux MCG data made by the study reader(s) will not be known to the patient's treating physician. Similarly, the patient's coronary physiology data, diagnosis, or interventions made by the patient's treating physician in following the standard of care will not be known to any of the scan readers. Except for the introduction of the MCG scan, there will be no other alteration to the patient standard of care.

ELIGIBILITY:
INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all the following criteria:

1. ≥ 18 years of age at the time of enrollment.
2. Willing to provide written informed consent.
3. Signs and symptoms of chest pain prompted further evaluation by a coronary angiogram within the previous 5 years.
4. Invasive CFR (via bolus thermodilution) completed within 180 days, or scheduled within 30 days, of informed consent.

   4.1. CFR must be performed in the mid Left Anterior Descending (LAD) vessel.
5. Successfully passing CardioFlux MCG Quality Preview prior to MCG study scan. 5.1. Patients must be able to fit into the device. 5.2. Patients must be able to lie supine for 5 minutes. 5.3. Patients must not have any of the following: 5.3.1. Presence of ferromagnetic metal between the sternal notch and costal margin of the rib cage.

5.3.2. Implanted pacemakers or cardioverter/defibrillators. 5.3.3. Implanted infusion pumps and/or neuro stimulators. 5.3.4. Note: sternotomy wires and stents are acceptable. 5.3.5. Note: Failure to meet inclusion criteria 5.3 will render the MCG scan uninterpretable. However, any patient who may be scanned with the presence of any of the above objects is not at any risk of harm by the device. Prosthetic joints are allowed if the MCG Quality Preview is acceptable.

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Obstructive CAD (either anatomical or physiological) defined as:

   1.1. ≥ 70% lesion in any major epicardial or branch vessel by CT or invasive Angiography; 1.2. ≥ 50% lesion in the Left Main (LM) vessel by CT or invasive Angiography; 1.3. or either an FFR<0.80 or iFR or RFR <0.89 in the obstructed vessel,
2. Any of the following cardiac pathologies:

   2.1. Epicardial spasm. 2.2. History of non-ischemic dilated or hypertrophic cardiomyopathy. 2.3. Suspected myocarditis. 2.4. Documented acute coronary syndrome (ACS) within previous 30 days. 2.5. Known left ventricular ejection fraction (LVEF) <45% on most recent assessment (can be via ECHO), or hospitalization for Reduced ejection fraction within 180 days. (HFpEF is allowed).

   2.6. Currently in atrial fibrillation or atrial flutter at the time of enrollment.

   2.7. Complete Bundle Branch Block. 2.8. Known moderate or severe valvular disease (anything besides mild). 2.9. Known severe Left ventricular hypertrophy (LVH) as determined by Echocardiography.

   2.10. Dextrocardia.
3. Known estimated glomerular filtration rate (eGFR) <30 ml/min.
4. Life expectancy <3-yrs. due to non-cardiovascular comorbidity.
5. Concurrent enrollment in a clinical trial in which therapeutic intervention is administered within 30 days of enrollment.
6. Prior enrollment in MICRO 1.0 and/or MICRO(T) data development study.
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 years and older with chronic/stable angina and no obstructive coronary artery disease (suspected INOCA) with completed invasive CFR measurement within 180 days or are scheduled to undergo invasive angiography with CFR assessment by bolus thermodilution within 30 days of informed consent at an enrolling clinical trial center.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CardioFlux MCG in determining the presence of CMD | 6 months
  Diagnostic accuracy of CardioFlux MCG in determining the presence of coronary microvascular dysfunction, as measured by AUC with ground truth defined as an invasive CFR <2.5 for bolus thermodilution method.
  H0: AUC<0.55 Ha: AUC≥0.55

SECONDARY OUTCOMES:
Sensitivity and specificity in determining presence of CMD (Rule In) | 6 months
  Patients who have confirmed presence of CMD via invasive CFR: Sensitivity and specificity of CardioFlux MCG in determining the presence of CMD with the gold standard defined as an invasive CFR <2.5 for thermodilution method as determined by a positive MCG scan output as defined by a Magnetic Dispersion Dynamics (MDD) score less than 41 fT/ms.
  Sensitivity
  * H0<0.30
  * Ha≥0.30
  Specificity
  * H0<0.70
  * Ha ≥0.70
Sensitivity and specificity in determining presence of CMD (Rule Out) | 6 months
  Patients who have confirmed absence of CMD via invasive CFR:
  Sensitivity
  * H0<0.70
  * Ha≥0.70
  Specificity
  * H0<0.30
  * Ha ≥0.30
ROC/AUC, sensitivity and specificity at CFR cut-offs of <2.0 and 3.0. | 6 months
  ROC/AUC, sensitivity and specificity for invasive CFR by thermodilution methods at CFR cut-offs of <2.0 and 3.0.
Patient-Reported Experiences with CardioFlux | 6 months
  Self-reported questionnaire (5 questions scored 1 (very dissatisfied) to 5 (very satisfied) with a minimum score of 5 and a maximum score of 25.
Participant Age | 6 months
  Age (years)
Participant Height | 6 months
  in meters; if known
Participant Weight | 6 months
  in kilograms; if known
Participant Gender at Birth | 6 months
  Male/Female
Index of Microvascular Resistance (IMR) | 6 months
  Sensitivity, Specificity, and ROC/AUC for CardioFlux will also be calculated against Index of Microvascular Resistance (IMR), defined as >25.
Comparison of bolus vs. continuous thermodilution | 6 months
  Comparison of bolus thermodilution (CFR-bolus) and continuous thermodilution (CFR-cont) against MCG when CFR-cont is available.
Number of Adverse Events | 6 months
  Safety will be monitored by the reporting of adverse events (related and non-related to the device) throughout the trial.

OTHER OUTCOMES:
Seattle Angina Questionnaire - 7 | 30 days
  For patients whose CFR was completed within 30 days of MCG scan, SAQ-7 scores may be measured and analyzed.
Comparison of functional vs structural CMD | 6 months
  Comparison of functional vs structural CMD will be analyzed (endothelial dependent vs independent).

CONTACTS AND LOCATIONS:
Overall Officials: Zoe E Swann, PhD, Study Director — Genetesis Inc.
Locations (8):
- United States (8):
  - University of Florida, Division of Cardiovascular Medicine, Gainesville, Florida
  - Saint Elizabeth Medical Center, Edgewood, Kentucky
  - Ascension St. John Hospital, Detroit, Michigan
  - Mayo Clinic, Cardiovascular Research, Rochester, Minnesota
  - St. Luke's Health System, Cardiovascular Research, Kansas City, Missouri
  - Hackensack Meridian Mountainside Medical Center, Montclair, New Jersey
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cardiovascular Medicine Research, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No